CLINICAL TRIAL: NCT00231413
Title: A Dose-range Study to Assess the Safety and Immunogenicity of a Novel HPV Vaccine When Administered Intramuscularly According to a 3-dose Schedule (0,1,6-month) in Healthy Adult Females (18-25 Years of Age)
Brief Title: Human Papilloma Virus Vaccine Immunogenicity and Safety Trial in Young Adult Women With GSK Bio's Novel HPV Vaccine.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 102115; 2004-003766-14 (EudraCT Number)
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Results first posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-11

CONDITIONS: Infections, Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This study was performed in a double-blinded manner. Blinding was maintained for all subjects and investigators and their study staff participating in this study with regard to the individual subject treatment (vaccine treatment) assignments allocated in this study.
  GSK personnel directly involved in the conduct of this study were also blinded to the subjects' treatment assignments.

ARMS (7):
- HPV-16/18 Group (Active Comparator): Female subjects who received 3 doses of the HPV-16/18 L1 AS04 vaccine intramuscularly, into the deltoid of the non-dominant arm according to a 3-dose 0, 1, 6-month vaccination schedule.
  Interventions: Biological: HPV 16/18 L1 AS04
- HPV-TETRA A Group (Experimental): Female subjects who received 3 doses of the HPV-16/18/31/45 L1/AS04 vaccine, formulation 1 intramuscularly, into the deltoid of the non-dominant arm according to a 3-dose 0, 1, 6-month vaccination schedule.
  Interventions: Biological: HPV-16/18/31/45 L1 AS04 Formulation 1
- HPV-TETRA B Group (Experimental): Female subjects who received 3 doses of the HPV-16/18/31/45 L1/AS04 vaccine, formulation 2 intramuscularly, into the deltoid of the non-dominant arm according to a 3-dose 0, 1, 6-month vaccination schedule.
  Interventions: Biological: HPV-16/18/31/45 L1 AS04 Formulation 2
- HPV-TETRA C Group (Experimental): Female subjects who received 3 doses of the HPV-16/18/31/45 L1/AS04 vaccine, formulation 3 intramuscularly, into the deltoid of the non-dominant arm according to a 3-dose 0, 1, 6-month vaccination schedule.
  Interventions: Biological: HPV-16/18/31/45 L1 AS04 Formulation 3
- HPV-TETRA D Group (Experimental): Female subjects who received 3 doses of the HPV-16/18/31/45 L1/AS04 vaccine, formulation 4 intramuscularly, into the deltoid of the non-dominant arm according to a 3-dose 0, 1, 6-month vaccination schedule.
  Interventions: Biological: HPV-16/18/31/45 L1 AS04 Formulation 4
- HPV-TETRA E Group (Experimental): Female subjects who received 3 doses of the HPV-16/18/31/45 L1/AS04 vaccine, formulation 5 intramuscularly, into the deltoid of the non-dominant arm according to a 3-dose 0, 1, 6-month vaccination schedule.
  Interventions: Biological: HPV-16/18/31/45 L1 AS04 Formulation 5
- HPV-TETRA F Group (Experimental): Female subjects who received 3 doses of the HPV-16/18/31/45 L1/AS04 vaccine, formulation 6 intramuscularly, into the deltoid of the non-dominant arm according to a 3-dose 0, 1, 6-month vaccination schedule.
  Interventions: Biological: HPV-16/18/31/45 L1 AS04 Formulation 6

INTERVENTIONS:
Biological: HPV 16/18 L1 AS04 — 3 doses of 0.6 mL supplied as a liquid in individual pre-filled syringes administered intramuscularly in the deltoid muscle of the non-dominant arm, at Day 0, Month 1 and Month 6.
  Arms: HPV-16/18 Group
Biological: HPV-16/18/31/45 L1 AS04 Formulation 1 — 3 doses of 0.6 mL supplied as a liquid in individual pre-filled syringes administered intramuscularly in the deltoid muscle of the non-dominant arm, at Day 0, Month 1 and Month 6.
  Arms: HPV-TETRA A Group
Biological: HPV-16/18/31/45 L1 AS04 Formulation 2 — 3 doses of 0.6 mL supplied as a liquid in individual pre-filled syringes administered intramuscularly in the deltoid muscle of the non-dominant arm, at Day 0, Month 1 and Month 6.
  Arms: HPV-TETRA B Group
Biological: HPV-16/18/31/45 L1 AS04 Formulation 3 — 3 doses of 0.6 mL supplied as a liquid in individual pre-filled syringes administered intramuscularly in the deltoid muscle of the non-dominant arm, at Day 0, Month 1 and Month 6.
  Arms: HPV-TETRA C Group
Biological: HPV-16/18/31/45 L1 AS04 Formulation 4 — 3 doses of 0.6 mL supplied as a liquid in individual pre-filled syringes administered intramuscularly in the deltoid muscle of the non-dominant arm, at Day 0, Month 1 and Month 6.
  Arms: HPV-TETRA D Group
Biological: HPV-16/18/31/45 L1 AS04 Formulation 5 — 3 doses of 0.6 mL supplied as a liquid in individual pre-filled syringes administered intramuscularly in the deltoid muscle of the non-dominant arm, at Day 0, Month 1 and Month 6.
  Arms: HPV-TETRA E Group
Biological: HPV-16/18/31/45 L1 AS04 Formulation 6 — 3 doses of 0.6 mL supplied as a liquid in individual pre-filled syringes administered intramuscularly in the deltoid muscle of the non-dominant arm, at Day 0, Month 1 and Month 6.
  Arms: HPV-TETRA F Group

SUMMARY:
Human Papilloma viruses (HPV) are viruses that cause infections of the skin and genitals in men and women. Several types of HPV infection are transmitted by sexual activity and, in women, can infect the cervix (part of the uterus or womb). This infection, if it persists, can lead over a long period of time to cancer of the cervix in women. In collaboration with MedImmune Inc., GlaxoSmithKline Biologicals has developed a HPV vaccine against the oncogenic types HPV-16 and HPV-18 formulated with the adjuvant AS04. GSK Biologicals is also evaluating novel HPV vaccine formulations.This study will evaluate the immunogenicity and safety of a novel GSK Biologicals HPV vaccine in women 18-25 years of age at study start. Approximately 376 study subjects will receive the novel HPV vaccine or the control vaccine administered intramuscularly according to a 0-1-6 month schedule.

ELIGIBILITY:
Inclusion Criteria:

* A woman between, and including, 18 and 25 years of age at the time of the first vaccination
* Written informed consent from the subject prior to enrolment
* Subject must be free of obvious health problems
* Subject must be of non-childbearing potential and have had no more than 6 lifetime sexual partners

Exclusion Criteria:

* Pregnant or breastfeeding
* A woman planning to become pregnant or planning to discontinue contraceptive precautions during approximately the first nine months of the study (Month 0-8)
* Known acute or chronic, clinically significant pulmonary, cardiovascular, neurologic, hepatic or renal functional abnormality
* History of chronic condition(s) requiring treatment such as cancer, chronic hepatitis or kidney disease(s), diabetes, or autoimmune disease
* Previous vaccination against human papillomavirus (HPV)

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 383 (Actual)
Dates: Start 2005-03-04 (Actual); Primary Completion 2006-03-27 (Actual); Study Completion 2006-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (4):
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Kingston, Rhode Island
  - GSK Investigational Site, Salt Lake City, Utah
- Belgium (6):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Roeselare
  - GSK Investigational Site, Wilrijk

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below).
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=1504

REFERENCES:
- [Background] Van Damme P, Leroux-Roels G, Simon P, Foidart JM, Donders G, Hoppenbrouwers K, Levin M, Tibaldi F, Poncelet S, Moris P, Dessy F, Giannini SL, Descamps D, Dubin G. Effects of varying antigens and adjuvant systems on the immunogenicity and safety of investigational tetravalent human oncogenic papillomavirus vaccines: results from two randomized trials. Vaccine. 2014 Jun 17;32(29):3694-705. doi: 10.1016/j.vaccine.2014.03.040. Epub 2014 Mar 25. PMID 24674663
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 102115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 102115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 102115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 102115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 102115 are summarised with studies 107919 and 108052 on the GSK Clinical Study Register.
- Available data/document: Informed Consent Form: 102115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 102115 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Started | 88 | 50 | 49 | 48 | 48 | 50 | 50
Completed | 80 | 45 | 42 | 45 | 45 | 45 | 46
Not Completed | 8 | 5 | 7 | 3 | 3 | 5 | 4
Not completed — Non-serious AE | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1 | 4 | 2 | 2 | 0 | 3
Not completed — Migrated/moved from study area | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 4 | 4 | 1 | 1 | 1 | 4 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group | Total
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50 | 383
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.9 (2.03) | 21.5 (2.18) | 21.2 (2.07) | 21.1 (2.09) | 21.4 (2.27) | 21.2 (2.26) | 20.7 (1.91) | 21.1 (2.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 50 | 49 | 48 | 48 | 50 | 50 | 383
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 6
  White/caucasian | 80 | 50 | 46 | 46 | 42 | 44 | 47 | 355
  Arabic/north african | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  East/south east asian | 4 | 0 | 0 | 0 | 2 | 0 | 0 | 6
  South asian | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 3
  American hispanic | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 5
  Japanese | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Other, not specified | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Anti-Human Papillomavirus (Anti-HPV)-16 at Month 7
Description: Seroconversion was defined as the appearance of anti-HPV-16 antibodies [i.e. antibody titer greater than or equal to (≥) the cut-off value] in the serum of subjects seronegative before vaccination. The cut-off value was 8 enzyme-linked immunosorbent assay (ELISA) units per milliliter (EL.U/mL).
Time Frame: At Month 7
Population: The analysis was based on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects with available data concerning immunogenicity outcome measures, seronegative before vaccination and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 62 | 32 | 31 | 23 | 33 | 28 | 33
Participants | 62 | 27 | 31 | 23 | 33 | 28 | 33

2. Primary Outcome: Number of Seroconverted Subjects for Anti-HPV-18 at Month 7
Description: Seroconversion was defined as the appearance of anti-HPV-18 antibodies (i.e. antibody titer ≥ cut-off value) in the serum of subjects seronegative before vaccination. The cut-off value was 7 EL.U/mL.
Time Frame: At Month 7
Population: The analysis was based on the ATP cohort for immunogenicity, which included all evaluable subjects with available data concerning immunogenicity outcome measures, who were seronegative before vaccination and for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 59 | 30 | 37 | 34 | 27 | 33 | 36
Participants | 59 | 30 | 37 | 34 | 27 | 33 | 36

3. Primary Outcome: Anti-HPV-16 Antibody Titers Assessed by ELISA at Month 7
Description: Anti-HPV-16 antibody titers were presented as Geometric Mean Titers (GMT) and expressed in EL.U/mL.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 62 | 27 | 31 | 23 | 33 | 28 | 33
EL.U/mL | 9086.1 [7231.1 to 11417.1] | 5757.4 [4283.9 to 7737.8] | 7897.7 [5825.2 to 10707.6] | 7524.1 [5678.1 to 9970.2] | 5986.4 [4485.2 to 7990.2] | 8483.5 [6257.6 to 11501.1] | 7605.0 [5818.7 to 9939.6]

4. Primary Outcome: Anti-HPV-18 Antibody Titers Assessed by ELISA at Month 7
Description: Anti-HPV-18 antibody titers were presented as Geometric Mean Titers and expressed in EL.U/mL.
Time Frame: At Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 59 | 30 | 37 | 34 | 27 | 33 | 36
EL.U/mL | 5184.5 [4211.1 to 6382.8] | 3061.3 [2231.7 to 4199.4] | 3640.2 [2590.4 to 5115.6] | 3268.6 [2650.4 to 4031.1] | 2998.5 [2109.5 to 4262.1] | 3296.2 [2402.8 to 4521.8] | 3056.0 [2364.5 to 3949.5]

5. Secondary Outcome: Number of Seroconverted Subjects for Anti-HPV-16 at Month 2
Description: Seroconversion was defined as the appearance of anti-HPV-16 antibodies (i.e. antibody titer ≥ cut-off value) in the serum of subjects seronegative before vaccination. The cut-off value was 8 EL.U/mL.
Time Frame: At Month 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 62 | 27 | 31 | 23 | 33 | 28 | 33
Participants | 62 | 27 | 31 | 23 | 33 | 28 | 33

6. Secondary Outcome: Number of Seroconverted Subjects for Anti-HPV-18 at Month 2
Description: as for outcome 2
Time Frame: At Month 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 59 | 30 | 37 | 34 | 27 | 33 | 36
Participants | 59 | 30 | 37 | 34 | 27 | 33 | 36

7. Secondary Outcome: Anti-HPV-16 Antibody Titers Assessed by ELISA at Month 2
Description: Anti-HPV-16 antibody titers were presented as Geometric Mean Titers and expressed in EL.U/mL.
Time Frame: At Month 2
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 62 | 27 | 31 | 23 | 33 | 28 | 33
EL.U/mL | 3256.7 [2613.6 to 4058.0] | 2718.9 [2207.9 to 3348.1] | 2779.4 [2139.2 to 3611.2] | 2915.5 [2346.9 to 3621.9] | 2353.5 [1782.0 to 3108.2] | 3202.3 [2539.5 to 4038.0] | 2720.9 [2226.8 to 3324.6]

8. Secondary Outcome: Anti-HPV-18 Antibody Titers Assessed by ELISA at Month 2
Description: Anti-HPV-18 antibody titers were presented as Geometric Mean Titers and expressed in EL.U/mL.
Time Frame: At Month 2
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 59 | 30 | 37 | 34 | 27 | 33 | 36
EL.U/mL | 2530.1 [2007.0 to 3189.5] | 1731.5 [1311.6 to 2285.9] | 1875.9 [1464.0 to 2403.7] | 2082.2 [1682.3 to 2577.2] | 2048.8 [1566.9 to 2678.8] | 2003.1 [1575.4 to 2547.0] | 1820.0 [1412.2 to 2345.6]

9. Secondary Outcome: Number of Seroconverted Subjects for Anti-HPV-31 at Months 2 and 7
Description: Seroconversion was defined as the appearance of anti-HPV-31 antibodies (i.e. antibody titer ≥ cut-off value) in the serum of subjects seronegative before vaccination. The cut-off value was 59 EL.U/mL.
Time Frame: At Month 2 and Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 61 | 32 | 37 | 29 | 31 | 30 | 36
Participants
  Month 2: number analyzed (Participants) | 60 | 32 | 37 | 29 | 31 | 30 | 36
  Month 2 | 54 | 32 | 37 | 29 | 31 | 30 | 36
  Month 7 | 61 | 32 | 37 | 29 | 31 | 30 | 36

10. Secondary Outcome: Number of Seroconverted Subjects for Anti-HPV-45 at Months 2 and 7
Description: Seroconversion was defined as the appearance of anti-HPV-45 antibodies (i.e. antibody titer ≥ cut-off value) in the serum of subjects seronegative before vaccination. The cut-off value was 59 EL.U/mL.
Time Frame: At Month 2 and Month 7
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 56 | 33 | 31 | 27 | 32 | 34 | 35
Participants
  Month 2: number analyzed (Participants) | 55 | 33 | 31 | 27 | 32 | 34 | 35
  Month 2 | 54 | 33 | 31 | 27 | 32 | 34 | 35
  Month 7 | 56 | 33 | 31 | 27 | 32 | 34 | 35

11. Secondary Outcome: Anti-HPV-31 Antibody Titers Assessed by ELISA at Months 2 and 7
Description: Anti-HPV-31 antibody titers were presented as Geometric Mean Titers and expressed in EL.U/mL.
Time Frame: At Month 2 and Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 61 | 32 | 37 | 29 | 31 | 30 | 36
EL.U/mL
  Month 2: number analyzed (Participants) | 60 | 32 | 37 | 29 | 31 | 30 | 36
  Month 2 | 232.8 [178.0 to 304.5] | 3694.6 [2720.2 to 5018.0] | 6271.3 [4762.4 to 8258.3] | 4570.7 [3636.0 to 5745.6] | 5114.8 [3967.7 to 6593.5] | 4846.7 [3817.6 to 6153.3] | 5627.6 [4650.8 to 6809.6]
  Month 7 | 920.5 [705.8 to 1200.6] | 7909.0 [5712.3 to 10950.4] | 14957.8 [11096.1 to 20163.5] | 9688.5 [7660.9 to 12252.7] | 11768.3 [8598.0 to 16107.6] | 9139.9 [6334.9 to 13186.9] | 12652.0 [10052.5 to 15923.6]

12. Secondary Outcome: Anti-HPV-45 Antibody Titers Assessed by ELISA at Months 2 and 7
Description: Anti-HPV-45 antibody titers were presented as Geometric Mean Titers and expressed in EL.U/mL.
Time Frame: At Month 2 and Month 7
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 56 | 33 | 31 | 27 | 32 | 34 | 35
EL.U/mL
  Month 2: number analyzed (Participants) | 55 | 33 | 31 | 27 | 32 | 34 | 35
  Month 2 | 317.4 [246.2 to 409.2] | 1550.7 [1158.1 to 2076.5] | 2613.9 [1980.7 to 3449.5] | 1893.7 [1513.2 to 2369.8] | 2113.3 [1602.9 to 2786.4] | 2217.4 [1763.8 to 2787.7] | 2208.9 [1718.5 to 2839.4]
  Month 7 | 915.7 [732.1 to 1145.3] | 4719.4 [3631.1 to 6133.9] | 7923.1 [5902.7 to 10635.0] | 5851.8 [4400.7 to 7781.4] | 6027.6 [4463.6 to 8139.4] | 6266.4 [4514.6 to 8698.1] | 6149.5 [4805.2 to 7869.8]

13. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any solicited local symptom regardless of their intensity grade. Grade 3 pain = significant pain at rest, that prevented normal every day activity. Grade 3 redness/swelling = redness/swelling above 50 millimeters (mm). All the reported local symptoms are considered related to the vaccination in the study.
Time Frame: During the 7 day post-vaccination period following each dose and across doses
Population: The analysis was based on the Total Vaccinated Cohort (TVC), which included all subjects with at least one vaccine administration documented, for whom data were available at the specified time point and had symptom sheets completed.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 86 | 49 | 47 | 46 | 46 | 50 | 48
Participants
  Any Pain - Dose 1 | 81 | 45 | 44 | 45 | 44 | 49 | 46
  Grade 3 Pain - Dose 1 | 6 | 6 | 5 | 6 | 5 | 5 | 7
  Any Pain - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Any Pain - Dose 2 | 70 | 42 | 40 | 42 | 40 | 43 | 45
  Grade 3 Pain - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Grade 3 Pain - Dose 2 | 2 | 3 | 3 | 4 | 4 | 4 | 3
  Any Pain - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Any Pain - Dose 3 | 68 | 40 | 33 | 40 | 37 | 40 | 39
  Grade 3 Pain - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Grade 3 Pain - Dose 3 | 7 | 6 | 3 | 10 | 7 | 6 | 7
  Any Pain - Across doses | 81 | 48 | 46 | 45 | 44 | 50 | 47
  Grade 3 Pain - Across doses | 10 | 12 | 7 | 14 | 11 | 12 | 12
  Any Redness - Dose 1 | 20 | 10 | 8 | 12 | 15 | 18 | 11
  Grade 3 Redness - Dose 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Any Redness - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Any Redness - Dose 2 | 21 | 18 | 9 | 10 | 14 | 15 | 13
  Grade 3 Redness - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Grade 3 Redness - Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Redness - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Any Redness - Dose 3 | 22 | 17 | 12 | 15 | 13 | 13 | 13
  Grade 3 Redness - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Grade 3 Redness - Dose 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Any Redness - Across doses | 36 | 28 | 15 | 22 | 24 | 22 | 25
  Grade 3 Redness - Across doses | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Any Swelling - Dose 1 | 17 | 10 | 6 | 8 | 6 | 14 | 9
  Grade 3 Swelling - Dose 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Any Swelling - Dose 2 | 17 | 11 | 3 | 6 | 16 | 18 | 6
  Grade 3 Swelling - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Grade 3 Swelling - Dose 2 | 1 | 0 | 0 | 0 | 2 | 2 | 0
  Any Swelling - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Any Swelling - Dose 3 | 23 | 14 | 8 | 11 | 15 | 16 | 11
  Grade 3 Swelling - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Grade 3 Swelling - Dose 3 | 1 | 0 | 0 | 1 | 1 | 1 | 0
  Any Swelling - Across doses | 33 | 22 | 12 | 18 | 21 | 27 | 19
  Grade 3 Swelling - Across doses | 2 | 0 | 0 | 1 | 2 | 2 | 0

14. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, fever, gastrointestinal symptoms, headache, myalgia, rash and urticaria. Any = occurrence of any solicited general symptom regardless of intensity grade or relationship to vaccination. Any Fever = axillary temperature greater than or equal to (≥) 37.5 degrees Celsius (°C). Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever greater than (>) 39.0°C. Related = general symptom assessed by the investigator as causally related to the vaccination.
Time Frame: During the 7 day post-vaccination period following each dose and across doses
Population: The analysis was based on the TVC, which included all subjects with at least one vaccine administration documented, for whom data were available at the specified time point and had symptom sheets completed.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 86 | 49 | 47 | 46 | 46 | 50 | 48
Participants
  Any Artharlgia - Dose 1 | 6 | 6 | 4 | 6 | 10 | 5 | 4
  Grade 3 Arthralgia - Dose 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
  Related Arthralgia - Dose 1 | 2 | 5 | 2 | 4 | 7 | 3 | 4
  Any Artharlgia - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Any Artharlgia - Dose 2 | 4 | 11 | 3 | 4 | 2 | 3 | 5
  Grade 3 Arthralgia - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Grade 3 Arthralgia - Dose 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Related Arthralgia - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Related Arthralgia - Dose 2 | 2 | 10 | 3 | 2 | 1 | 1 | 4
  Any Artharlgia - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Any Artharlgia - Dose 3 | 3 | 4 | 7 | 4 | 2 | 3 | 7
  Grade 3 Arthralgia - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Grade 3 Arthralgia - Dose 3 | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Related Arthralgia - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Related Arthralgia - Dose 3 | 2 | 3 | 5 | 4 | 2 | 2 | 5
  Any Artharlgia - Across doses | 11 | 13 | 9 | 11 | 11 | 9 | 11
  Grade 3 Arthralgia - Across doses | 2 | 0 | 2 | 0 | 3 | 1 | 0
  Related Arthralgia - Across doses | 5 | 12 | 7 | 9 | 9 | 5 | 9
  Any Fatigue - Dose 1 | 37 | 23 | 24 | 19 | 20 | 27 | 25
  Grade 3 Fatigue - Dose 1 | 0 | 2 | 2 | 1 | 1 | 2 | 2
  Related Fatigue - Dose 1 | 26 | 13 | 16 | 8 | 15 | 22 | 20
  Any Fatigue - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Any Fatigue - Dose 2 | 32 | 19 | 13 | 18 | 19 | 21 | 16
  Grade 3 Fatigue - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Grade 3 Fatigue - Dose 2 | 1 | 2 | 3 | 2 | 3 | 1 | 0
  Related Fatigue - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Related Fatigue - Dose 2 | 22 | 14 | 10 | 10 | 14 | 16 | 11
  Any Fatigue - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Any Fatigue - Dose 3 | 28 | 16 | 15 | 18 | 14 | 22 | 20
  Grade 3 Fatigue - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Grade 3 Fatigue - Dose 3 | 0 | 1 | 1 | 1 | 3 | 2 | 1
  Related Fatigue - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Related Fatigue - Dose 3 | 18 | 15 | 11 | 14 | 12 | 16 | 14
  Any Fatigue - Across doses | 54 | 33 | 30 | 32 | 25 | 34 | 31
  Grade 3 Fatigue - Across doses | 1 | 4 | 6 | 3 | 5 | 5 | 3
  Related Fatigue - Across doses | 42 | 28 | 24 | 22 | 22 | 27 | 27
  Any Fever - Dose 1 | 4 | 2 | 2 | 1 | 4 | 1 | 1
  Grade 3 Fever - Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever - Dose 1 | 2 | 2 | 0 | 1 | 3 | 0 | 1
  Any Fever - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Any Fever - Dose 2 | 2 | 2 | 2 | 3 | 3 | 2 | 1
  Grade 3 Fever - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Grade 3 Fever - Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Related Fever - Dose 2 | 1 | 2 | 1 | 2 | 3 | 1 | 1
  Any Fever - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Any Fever - Dose 3 | 7 | 1 | 1 | 1 | 4 | 1 | 1
  Grade 3 Fever - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Grade 3 Fever - Dose 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Related Fever - Dose 3 | 3 | 1 | 0 | 1 | 4 | 1 | 1
  Any Fever - Across doses | 10 | 4 | 4 | 3 | 9 | 4 | 2
  Grade 3 Fever - Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever - Across doses | 5 | 4 | 1 | 3 | 9 | 2 | 2
  Any Gastrointestinal - Dose 1 | 25 | 10 | 13 | 10 | 9 | 10 | 13
  Grade 3 Gastrointestinal - Dose 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
  Related Gastrointestinal - Dose 1 | 14 | 4 | 6 | 3 | 8 | 5 | 7
  Any Gastrointestinal - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Any Gastrointestinal - Dose 2 | 16 | 10 | 8 | 6 | 6 | 10 | 4
  Grade 3 Gastrointestinal - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Grade 3 Gastrointestinal - Dose 2 | 1 | 1 | 1 | 0 | 2 | 0 | 0
  Related Gastrointestinal - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Related Gastrointestinal - Dose 2 | 7 | 6 | 4 | 1 | 3 | 8 | 2
  Any Gastrointestinal - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Any Gastrointestinal - Dose 3 | 17 | 5 | 7 | 6 | 8 | 7 | 6
  Grade 3 Gastrointestinal - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Grade 3 Gastrointestinal - Dose 3 | 2 | 0 | 0 | 2 | 1 | 1 | 0
  Related Gastrointestinal - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Related Gastrointestinal - Dose 3 | 5 | 1 | 5 | 4 | 4 | 2 | 4
  Any Gastrointestinal - Across doses | 36 | 15 | 18 | 20 | 17 | 17 | 18
  Grade 3 Gastrointestinal - Across doses | 4 | 1 | 2 | 2 | 2 | 1 | 1
  Related Gastrointestinal - Across doses | 18 | 8 | 12 | 8 | 10 | 10 | 11
  Any Headache - Dose 1 | 32 | 11 | 16 | 24 | 17 | 29 | 13
  Grade 3 Headache - Dose 1 | 2 | 1 | 0 | 1 | 1 | 1 | 1
  Related Headache - Dose 1 | 19 | 8 | 6 | 9 | 13 | 18 | 9
  Any Headache - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Any Headache - Dose 2 | 21 | 17 | 9 | 14 | 12 | 19 | 19
  Grade 3 Headache - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Grade 3 Headache - Dose 2 | 1 | 2 | 1 | 1 | 1 | 1 | 2
  Related Headache - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Related Headache - Dose 2 | 15 | 12 | 7 | 8 | 9 | 14 | 11
  Any Headache - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Any Headache - Dose 3 | 24 | 12 | 8 | 14 | 9 | 18 | 18
  Grade 3 Headache - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Grade 3 Headache - Dose 3 | 3 | 0 | 1 | 0 | 2 | 3 | 0
  Related Headache - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Related Headache - Dose 3 | 14 | 10 | 5 | 6 | 6 | 15 | 13
  Any Headache - Across doses | 45 | 24 | 23 | 31 | 22 | 33 | 27
  Grade 3 Headache - Across doses | 5 | 3 | 2 | 2 | 2 | 5 | 2
  Related Headache - Across doses | 32 | 17 | 15 | 16 | 19 | 25 | 21
  Any Myalgia - Dose 1 | 20 | 14 | 11 | 8 | 11 | 14 | 10
  Grade 3 Myalgia - Dose 1 | 0 | 1 | 3 | 4 | 0 | 1 | 1
  Related Myalgia - Dose 1 | 14 | 11 | 9 | 5 | 11 | 10 | 9
  Any Myalgia - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Any Myalgia - Dose 2 | 12 | 11 | 7 | 9 | 9 | 5 | 7
  Grade 3 Myalgia - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Grade 3 Myalgia - Dose 2 | 1 | 0 | 1 | 1 | 0 | 1 | 0
  Related Myalgia - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Related Myalgia - Dose 2 | 8 | 11 | 7 | 5 | 8 | 4 | 5
  Any Myalgia - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Any Myalgia - Dose 3 | 10 | 11 | 11 | 7 | 8 | 7 | 8
  Grade 3 Myalgia - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Grade 3 Myalgia - Dose 3 | 1 | 0 | 1 | 1 | 1 | 1 | 1
  Related Myalgia - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Related Myalgia - Dose 3 | 8 | 11 | 9 | 5 | 6 | 6 | 7
  Any Myalgia - Across doses | 25 | 18 | 19 | 16 | 17 | 19 | 15
  Grade 3 Myalgia - Across doses | 2 | 1 | 3 | 5 | 1 | 2 | 2
  Related Myalgia - Across doses | 20 | 16 | 16 | 13 | 15 | 14 | 13
  Any Rash - Dose 1 | 4 | 1 | 1 | 1 | 4 | 1 | 1
  Grade 3 Rash - Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Rash - Dose 1 | 0 | 0 | 0 | 0 | 3 | 1 | 1
  Any Rash - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Any Rash - Dose 2 | 3 | 2 | 1 | 0 | 0 | 3 | 0
  Grade 3 Rash - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Grade 3 Rash - Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Rash - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Related Rash - Dose 2 | 3 | 0 | 1 | 0 | 0 | 2 | 0
  Any Rash - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Any Rash - Dose 3 | 1 | 1 | 1 | 1 | 1 | 0 | 2
  Grade 3 Rash - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Grade 3 Rash - Dose 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Rash - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Related Rash - Dose 3 | 1 | 1 | 0 | 1 | 1 | 0 | 1
  Any Rash - Across doses | 6 | 4 | 2 | 2 | 4 | 3 | 2
  Grade 3 Rash - Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Rash - Across doses | 3 | 1 | 1 | 1 | 4 | 2 | 2
  Any Urticaria - Dose 1 | 1 | 1 | 3 | 0 | 0 | 1 | 2
  Grade 3 Urticaria - Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Urticaria - Dose 1 | 1 | 1 | 2 | 0 | 0 | 1 | 2
  Any Urticaria - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Any Urticaria - Dose 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Urticaria - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Grade 3 Urticaria - Dose 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Urticaria - Dose 2: number analyzed (Participants) | 82 | 46 | 42 | 45 | 45 | 49 | 47
  Related Urticaria - Dose 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Any Urticaria - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Any Urticaria - Dose 3 | 2 | 1 | 1 | 0 | 0 | 0 | 1
  Grade 3 Urticaria - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Grade 3 Urticaria - Dose 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Urticaria - Dose 3: number analyzed (Participants) | 79 | 44 | 42 | 43 | 44 | 44 | 46
  Related Urticaria - Dose 3 | 2 | 1 | 0 | 0 | 0 | 0 | 1
  Any Urticaria - Across doses | 3 | 2 | 3 | 0 | 0 | 1 | 3
  Grade 3 Urticaria - Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Urticaria - Across doses | 3 | 2 | 2 | 0 | 0 | 1 | 3

15. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited adverse event (AE) was defined as any AE reported in addition to those solicited during the clinical study. Also, any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event. Any is defined as the occurrence of any unsolicited AE irrespective of its intensity grade and relationship to vaccination. Grade 3 unsolicited AE = an AE that prevented normal, everyday activities. Related AE = an AE assessed by the investigator as causally related to the study vaccination.
Time Frame: During the 30-day post-vaccination period
Population: The analysis was based on the TVC, which included all subjects with at least one vaccine administration documented for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50
Participants
  Any AEs | 60 | 31 | 34 | 25 | 32 | 36 | 29
  Grade 3 AEs | 14 | 5 | 8 | 3 | 5 | 6 | 8
  Related AEs | 17 | 16 | 7 | 6 | 9 | 8 | 9

16. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity or were a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination.
Time Frame: From Day 0 to Month 7
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50
Participants | 1 | 2 | 0 | 2 | 1 | 0 | 0

17. Secondary Outcome: Number of Subjects With Any SAEs During the Extended Safety Follow-up
Description: as for outcome 16
Time Frame: From Day 0 to Month 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50
Participants | 2 | 2 | 1 | 3 | 2 | 0 | 0

18. Secondary Outcome: Number of Subjects Reporting Pregnancies and Outcomes of Reported Pregnancies
Description: Outcomes of reported pregnancies were: Healthy baby, Spontaneous abortion, Elective abortion.
Time Frame: From Day 0 to Month 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50
Participants
  Healthy baby | 0 | 0 | 2 | 1 | 0 | 1 | 2
  Spontaneous abortion | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Elective abortion | 1 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Subjects Reporting New Onset of Chronic Diseases (NOCDs)
Description: NOCDs assessed include chronic diseases such as autoimmune disorders, diabetes, allergies also asthma and pathognomic signs/symptoms of these diseases.
Time Frame: From Day 0 up to Month 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50
Participants | 5 | 1 | 6 | 1 | 3 | 1 | 2

20. Secondary Outcome: Number of Subjects Reporting Medically Significant Conditions
Description: Medically significant conditions are AEs prompting emergency room or physician visits that were not related to common diseases or routine visits for physical examination or vaccination, or SAEs that were not related to common diseases.
Time Frame: From Day 0 up to Month 12
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 88 | 50 | 49 | 48 | 48 | 50 | 50
Participants | 2 | 1 | 1 | 2 | 2 | 0 | 0

21. Secondary Outcome: Number of Subjects With Clinically Relevant Abnormalities in Biochemical and Haematological Parameters
Description: The parameters assessed were both biochemical (alanine aminotransferase = ALAT, creatinine = CREA, blood urea nitrogen = BUN) and haematological [basophils = BAS, eosinophils = EOS, red blood cells = RBC, hematocrit = HCT, hemoglobin = HGB, leukocytes (white blood cells) = WBC, lymphocytes = LYM, monocytes = MONO, neutrophils = NEU and platelets = PLA]. Abnormal values of a parameter at Months 2 and 7 are defined as below and above the normal ranges, as compared to the baseline status of the same parameter.
Time Frame: At Month 2 and Month 7
Population: The analysis was based on the TVC, which included all subjects with at least one vaccine administration documented for whom data were available at the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
Number analyzed (Participants) | 83 | 45 | 43 | 45 | 45 | 49 | 46
Participants
  ALAT, Normal (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 81 | 45 | 42 | 45 | 45 | 48 | 46
  ALAT, Normal (pre-vacc) - Normal (Month 2) | 78 | 43 | 42 | 44 | 42 | 47 | 46
  ALAT, Normal (pre-vacc) - Below (Month 2): number analyzed (Participants) | 81 | 45 | 42 | 45 | 45 | 48 | 46
  ALAT, Normal (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALAT, Normal (pre-vacc) - Above (Month 2): number analyzed (Participants) | 81 | 45 | 42 | 45 | 45 | 48 | 46
  ALAT, Normal (pre-vacc) - Above (Month 2) | 2 | 2 | 0 | 1 | 2 | 1 | 0
  ALAT, Normal (pre-vacc) - Missing (Month 2): number analyzed (Participants) | 81 | 45 | 42 | 45 | 45 | 48 | 46
  ALAT, Normal (pre-vacc) - Missing (Month 2) | 1 | 0 | 0 | 0 | 1 | 0 | 0
  ALAT, Normal (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 78 | 44 | 41 | 45 | 44 | 43 | 45
  ALAT, Normal (pre-vacc) - Normal (Month 7) | 78 | 44 | 40 | 44 | 41 | 41 | 45
  ALAT, Normal (pre-vacc) - Below (Month 7): number analyzed (Participants) | 78 | 44 | 41 | 45 | 44 | 43 | 45
  ALAT, Normal (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALAT, Normal (pre-vacc) - Above (Month 7): number analyzed (Participants) | 78 | 44 | 41 | 45 | 44 | 43 | 45
  ALAT, Normal (pre-vacc) - Above (Month 7) | 0 | 0 | 1 | 1 | 3 | 1 | 0
  ALAT, Normal (pre-vacc) - Missing (Month 7): number analyzed (Participants) | 78 | 44 | 41 | 45 | 44 | 43 | 45
  ALAT, Normal (pre-vacc) - Missing (Month 7) | 0 | 0 | 0 | 0 | 0 | 1 | 0
  ALAT, Above (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 2 | 1 | 1 | 0 | 1 | 2 | 0
  ALAT, Above (pre-vacc) - Normal (Month 2) | 2 | 1 | 1 | 0 | 0 | 2 | 0
  ALAT, Above (pre-vacc) - Below (Month 2): number analyzed (Participants) | 2 | 1 | 1 | 0 | 1 | 2 | 0
  ALAT, Above (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALAT, Above (pre-vacc) - Above (Month 2): number analyzed (Participants) | 2 | 1 | 1 | 0 | 1 | 2 | 0
  ALAT, Above (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  ALAT, Above (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 2 | 1 | 1 | 0 | 1 | 2 | 0
  ALAT, Above (pre-vacc) - Normal (Month 7) | 2 | 1 | 1 | 0 | 1 | 2 | 0
  ALAT, Above (pre-vacc) - Below (Month 7): number analyzed (Participants) | 2 | 1 | 1 | 0 | 1 | 2 | 0
  ALAT, Above (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALAT, Above (pre-vacc) - Above (Month 7): number analyzed (Participants) | 2 | 1 | 1 | 0 | 1 | 2 | 0
  ALAT, Above (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Normal (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 80 | 43 | 42 | 42 | 44 | 48 | 45
  BAS, Normal (pre-vacc) - Normal (Month 2) | 80 | 43 | 42 | 42 | 43 | 48 | 45
  BAS, Normal (pre-vacc) - Below (Month 2): number analyzed (Participants) | 80 | 43 | 42 | 42 | 44 | 48 | 45
  BAS, Normal (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Normal (pre-vacc) - Above (Month 2): number analyzed (Participants) | 80 | 43 | 42 | 42 | 44 | 48 | 45
  BAS, Normal (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Normal (pre-vacc) - Missing (Month 2): number analyzed (Participants) | 80 | 43 | 42 | 42 | 44 | 48 | 45
  BAS, Normal (pre-vacc) - Missing (Month 2) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  BAS, Normal (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 77 | 42 | 41 | 42 | 43 | 43 | 44
  BAS, Normal (pre-vacc) - Normal (Month 7) | 76 | 40 | 40 | 41 | 43 | 43 | 44
  BAS, Normal (pre-vacc) - Below (Month 7): number analyzed (Participants) | 77 | 42 | 41 | 42 | 43 | 43 | 44
  BAS, Normal (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  BAS, Normal (pre-vacc) - Above (Month 7): number analyzed (Participants) | 77 | 42 | 41 | 42 | 43 | 43 | 44
  BAS, Normal (pre-vacc) - Above (Month 7) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  BAS, Normal (pre-vacc) - Missing (Month 7): number analyzed (Participants) | 77 | 42 | 41 | 42 | 43 | 43 | 44
  BAS, Normal (pre-vacc) - Missing (Month 7) | 0 | 1 | 1 | 1 | 0 | 0 | 0
  CREA, Normal (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 79 | 45 | 43 | 44 | 44 | 49 | 46
  CREA, Normal (pre-vacc) - Normal (Month 2) | 78 | 43 | 42 | 43 | 43 | 47 | 43
  CREA, Normal (pre-vacc) - Below (Month 2): number analyzed (Participants) | 79 | 45 | 43 | 44 | 44 | 49 | 46
  CREA, Normal (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CREA, Normal (pre-vacc) - Above (Month 2): number analyzed (Participants) | 79 | 45 | 43 | 44 | 44 | 49 | 46
  CREA, Normal (pre-vacc) - Above (Month 2) | 1 | 2 | 1 | 1 | 0 | 2 | 3
  CREA, Normal (pre-vacc) - Missing (Month 2): number analyzed (Participants) | 79 | 45 | 43 | 44 | 44 | 49 | 46
  CREA, Normal (pre-vacc) - Missing (Month 2) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  CREA, Normal (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 76 | 44 | 42 | 44 | 43 | 44 | 45
  CREA, Normal (pre-vacc) - Normal (Month 7) | 73 | 43 | 42 | 43 | 41 | 44 | 43
  CREA, Normal (pre-vacc) - Below (Month 7): number analyzed (Participants) | 76 | 44 | 42 | 44 | 43 | 44 | 45
  CREA, Normal (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CREA, Normal (pre-vacc) - Above (Month 7): number analyzed (Participants) | 76 | 44 | 42 | 44 | 43 | 44 | 45
  CREA, Normal (pre-vacc) - Above (Month 7) | 3 | 1 | 0 | 1 | 2 | 0 | 2
  CREA, Above (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 4 | 1 | 0 | 1 | 2 | 1 | 0
  CREA, Above (pre-vacc) - Normal (Month 2) | 3 | 0 | 0 | 0 | 1 | 1 | 0
  CREA, Above (pre-vacc) - Below (Month 2): number analyzed (Participants) | 4 | 1 | 0 | 1 | 2 | 1 | 0
  CREA, Above (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CREA, Above (pre-vacc) - Above (Month 2): number analyzed (Participants) | 4 | 1 | 0 | 1 | 2 | 1 | 0
  CREA, Above (pre-vacc) - Above (Month 2) | 1 | 1 | 0 | 1 | 1 | 0 | 0
  CREA, Above (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 4 | 1 | 0 | 1 | 2 | 1 | 0
  CREA, Above (pre-vacc) - Normal (Month 7) | 3 | 0 | 0 | 0 | 1 | 1 | 0
  CREA, Above (pre-vacc) - Below (Month 7): number analyzed (Participants) | 4 | 1 | 0 | 1 | 2 | 1 | 0
  CREA, Above (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CREA, Above (pre-vacc) - Above (Month 7): number analyzed (Participants) | 4 | 1 | 0 | 1 | 2 | 1 | 0
  CREA, Above (pre-vacc) - Above (Month 7) | 1 | 1 | 0 | 1 | 1 | 0 | 0
  EOS, Normal (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 73 | 41 | 42 | 39 | 43 | 46 | 45
  EOS, Normal (pre-vacc) - Normal (Month 2) | 67 | 40 | 42 | 38 | 39 | 45 | 41
  EOS, Normal (pre-vacc) - Below (Month 2): number analyzed (Participants) | 73 | 41 | 42 | 39 | 43 | 46 | 45
  EOS, Normal (pre-vacc) - Below (Month 2) | 3 | 1 | 0 | 1 | 0 | 1 | 1
  EOS, Normal (pre-vacc) - Above (Month 2): number analyzed (Participants) | 73 | 41 | 42 | 39 | 43 | 46 | 45
  EOS, Normal (pre-vacc) - Above (Month 2) | 3 | 0 | 0 | 0 | 3 | 0 | 3
  EOS, Normal (pre-vacc) - Missing (Month 2): number analyzed (Participants) | 73 | 41 | 42 | 39 | 43 | 43 | 45
  EOS, Normal (pre-vacc) - Missing (Month 2) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  EOS, Normal (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 70 | 40 | 41 | 39 | 42 | 41 | 44
  EOS, Normal (pre-vacc) - Normal (Month 7) | 63 | 38 | 40 | 38 | 40 | 38 | 43
  EOS, Normal (pre-vacc) - Below (Month 7): number analyzed (Participants) | 70 | 40 | 41 | 39 | 42 | 41 | 44
  EOS, Normal (pre-vacc) - Below (Month 7) | 3 | 0 | 0 | 0 | 0 | 2 | 1
  EOS, Normal (pre-vacc) - Above (Month 7): number analyzed (Participants) | 70 | 40 | 41 | 39 | 42 | 41 | 44
  EOS, Normal (pre-vacc) - Above (Month 7) | 4 | 1 | 0 | 1 | 2 | 1 | 0
  EOS, Normal (pre-vacc) - Missing (Month 7): number analyzed (Participants) | 70 | 40 | 41 | 39 | 42 | 41 | 44
  EOS, Normal (pre-vacc) - Missing (Month 7) | 0 | 1 | 1 | 0 | 0 | 0 | 0
  EOS, Above (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 4 | 0 | 0 | 1 | 0 | 2 | 1
  EOS, Above (pre-vacc) - Normal (Month 2) | 4 | 0 | 0 | 0 | 0 | 2 | 0
  EOS, Above (pre-vacc) - Below (Month 2): number analyzed (Participants) | 4 | 0 | 0 | 1 | 0 | 0 | 1
  EOS, Above (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  EOS, Above (pre-vacc) - Above (Month 2): number analyzed (Participants) | 4 | 0 | 0 | 1 | 0 | 2 | 1
  EOS, Above (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 1 | 0 | 0 | 1
  EOS, Above (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 4 | 0 | 0 | 1 | 0 | 2 | 1
  EOS, Above (pre-vacc) - Normal (Month 7) | 4 | 0 | 0 | 0 | 0 | 1 | 0
  EOS, Above (pre-vacc) - Below (Month 7): number analyzed (Participants) | 4 | 0 | 0 | 1 | 0 | 2 | 1
  EOS, Above (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  EOS, Above (pre-vacc) - Above (Month 7): number analyzed (Participants) | 4 | 0 | 0 | 1 | 0 | 2 | 1
  EOS, Above (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 1 | 0 | 1 | 1
  EOS, Below (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 3 | 2 | 0 | 2 | 1 | 0 | 0
  EOS, Below (pre-vacc) - Normal (Month 2) | 3 | 1 | 0 | 2 | 1 | 0 | 0
  EOS, Below (pre-vacc) - Below (Month 2): number analyzed (Participants) | 3 | 2 | 0 | 2 | 1 | 0 | 0
  EOS, Below (pre-vacc) - Below (Month 2) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  EOS, Below (pre-vacc) - Above (Month 2): number analyzed (Participants) | 3 | 2 | 0 | 2 | 1 | 0 | 0
  EOS, Below (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  EOS, Below (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 3 | 2 | 0 | 2 | 1 | 0 | 0
  EOS, Below (pre-vacc) - Normal (Month 7) | 1 | 1 | 0 | 2 | 1 | 0 | 0
  EOS, Below (pre-vacc) - Below (Month 7): number analyzed (Participants) | 3 | 2 | 0 | 2 | 1 | 0 | 0
  EOS, Below (pre-vacc) - Below (Month 7) | 2 | 1 | 0 | 0 | 0 | 0 | 0
  EOS, Below (pre-vacc) - Above (Month 7): number analyzed (Participants) | 3 | 2 | 0 | 2 | 1 | 0 | 0
  EOS, Below (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HCT, Normal (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 75 | 41 | 41 | 40 | 43 | 49 | 42
  HCT, Normal (pre-vacc) - Normal (Month 2) | 73 | 39 | 41 | 40 | 39 | 45 | 41
  HCT, Normal (pre-vacc) - Below (Month 2): number analyzed (Participants) | 75 | 41 | 41 | 40 | 43 | 49 | 42
  HCT, Normal (pre-vacc) - Below (Month 2) | 0 | 2 | 0 | 0 | 1 | 2 | 0
  HCT, Normal (pre-vacc) - Above (Month 2): number analyzed (Participants) | 75 | 41 | 41 | 40 | 43 | 49 | 42
  HCT, Normal (pre-vacc) - Above (Month 2) | 2 | 0 | 0 | 0 | 2 | 2 | 1
  HCT, Normal (pre-vacc) - Missing (Month 2): number analyzed (Participants) | 75 | 41 | 41 | 40 | 43 | 49 | 42
  HCT, Normal (pre-vacc) - Missing (Month 2) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  HCT, Normal (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 72 | 41 | 40 | 40 | 42 | 44 | 41
  HCT, Normal (pre-vacc) - Normal (Month 7) | 71 | 38 | 40 | 40 | 41 | 43 | 39
  HCT, Normal (pre-vacc) - Below (Month 7): number analyzed (Participants) | 72 | 41 | 40 | 40 | 42 | 44 | 41
  HCT, Normal (pre-vacc) - Below (Month 7) | 1 | 2 | 0 | 0 | 0 | 1 | 0
  HCT, Normal (pre-vacc) - Above (Month 7): number analyzed (Participants) | 72 | 41 | 40 | 40 | 42 | 44 | 41
  HCT, Normal (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 0 | 1 | 0 | 2
  HCT, Normal (pre-vacc) - Missing (Month 7): number analyzed (Participants) | 72 | 41 | 40 | 40 | 42 | 44 | 41
  HCT, Normal (pre-vacc) - Missing (Month 7) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  HCT, Above (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 6 | 3 | 2 | 2 | 1 | 0 | 3
  HCT, Above (pre-vacc) - Normal (Month 2) | 4 | 2 | 2 | 2 | 1 | 0 | 2
  HCT, Above (pre-vacc) - Below (Month 2): number analyzed (Participants) | 6 | 3 | 2 | 2 | 1 | 0 | 3
  HCT, Above (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HCT, Above (pre-vacc) - Above (Month 2): number analyzed (Participants) | 6 | 3 | 2 | 2 | 1 | 0 | 3
  HCT, Above (pre-vacc) - Above (Month 2) | 2 | 1 | 0 | 0 | 0 | 0 | 1
  HCT, Above (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 6 | 3 | 2 | 2 | 1 | 0 | 3
  HCT, Above (pre-vacc) - Normal (Month 7) | 5 | 3 | 2 | 2 | 0 | 0 | 2
  HCT, Above (pre-vacc) - Below (Month 7): number analyzed (Participants) | 6 | 3 | 2 | 2 | 1 | 0 | 3
  HCT, Above (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HCT, Above (pre-vacc) - Above (Month 7): number analyzed (Participants) | 6 | 3 | 2 | 2 | 1 | 0 | 3
  HCT, Above (pre-vacc) - Above (Month 7) | 1 | 0 | 0 | 0 | 1 | 0 | 1
  HCT, Below (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 2 | 2 | 0 | 3 | 2 | 1 | 1
  HCT, Below (pre-vacc) - Normal (Month 2) | 1 | 2 | 0 | 3 | 2 | 0 | 1
  HCT, Below (pre-vacc) - Below (Month 2): number analyzed (Participants) | 2 | 2 | 0 | 3 | 2 | 1 | 1
  HCT, Below (pre-vacc) - Below (Month 2) | 1 | 0 | 0 | 0 | 0 | 1 | 0
  HCT, Below (pre-vacc) - Above (Month 2): number analyzed (Participants) | 2 | 2 | 0 | 3 | 2 | 1 | 1
  HCT, Below (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HCT, Below (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 2 | 1 | 0 | 3 | 2 | 1 | 1
  HCT, Below (pre-vacc) - Normal (Month 7) | 2 | 0 | 0 | 2 | 2 | 0 | 0
  HCT, Below (pre-vacc) - Below (Month 7): number analyzed (Participants) | 2 | 1 | 0 | 3 | 2 | 1 | 1
  HCT, Below (pre-vacc) - Below (Month 7) | 0 | 1 | 0 | 1 | 0 | 1 | 1
  HCT, Below (pre-vacc) - Above (Month 7): number analyzed (Participants) | 2 | 1 | 0 | 3 | 2 | 1 | 1
  HCT, Below (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYM, Normal (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 73 | 41 | 37 | 39 | 41 | 45 | 42
  LYM, Normal (pre-vacc) - Normal (Month 2) | 70 | 38 | 36 | 39 | 38 | 40 | 40
  LYM, Normal (pre-vacc) - Below (Month 2): number analyzed (Participants) | 73 | 41 | 37 | 39 | 41 | 41 | 42
  LYM, Normal (pre-vacc) - Below (Month 2) | 1 | 1 | 0 | 0 | 1 | 2 | 0
  LYM, Normal (pre-vacc) - Above (Month 2): number analyzed (Participants) | 73 | 41 | 37 | 39 | 41 | 41 | 42
  LYM, Normal (pre-vacc) - Above (Month 2) | 2 | 2 | 1 | 0 | 1 | 3 | 2
  LYM, Normal (pre-vacc) - Missing (Month 2): number analyzed (Participants) | 73 | 41 | 37 | 39 | 41 | 41 | 42
  LYM, Normal (pre-vacc) - Missing (Month 2) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  LYM, Normal (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 70 | 40 | 36 | 39 | 40 | 40 | 41
  LYM, Normal (pre-vacc) - Normal (Month 7) | 65 | 35 | 34 | 38 | 39 | 37 | 39
  LYM, Normal (pre-vacc) - Below (Month 7): number analyzed (Participants) | 70 | 40 | 36 | 39 | 40 | 40 | 41
  LYM, Normal (pre-vacc) - Below (Month 7) | 2 | 1 | 1 | 0 | 0 | 1 | 1
  LYM, Normal (pre-vacc) - Above (Month 7): number analyzed (Participants) | 70 | 40 | 36 | 39 | 40 | 40 | 41
  LYM, Normal (pre-vacc) - Above (Month 7) | 2 | 3 | 1 | 1 | 1 | 2 | 1
  LYM, Normal (pre-vacc) - Missing (Month 7): number analyzed (Participants) | 70 | 40 | 36 | 39 | 40 | 40 | 41
  LYM, Normal (pre-vacc) - Missing (Month 7) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  LYM, Above (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 5 | 1 | 4 | 2 | 2 | 2 | 1
  LYM, Above (pre-vacc) - Normal (Month 2) | 3 | 1 | 4 | 2 | 1 | 2 | 0
  LYM, Above (pre-vacc) - Below (Month 2): number analyzed (Participants) | 5 | 1 | 4 | 2 | 2 | 2 | 1
  LYM, Above (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYM, Above (pre-vacc) - Above (Month 2): number analyzed (Participants) | 5 | 1 | 4 | 2 | 2 | 2 | 1
  LYM, Above (pre-vacc) - Above (Month 2) | 2 | 0 | 0 | 0 | 1 | 0 | 1
  LYM, Above (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 5 | 1 | 4 | 2 | 2 | 2 | 1
  LYM, Above (pre-vacc) - Normal (Month 7) | 2 | 1 | 3 | 1 | 1 | 2 | 0
  LYM, Above (pre-vacc) - Below (Month 7): number analyzed (Participants) | 5 | 1 | 4 | 2 | 2 | 2 | 1
  LYM, Above (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYM, Above (pre-vacc) - Above (Month 7): number analyzed (Participants) | 5 | 1 | 4 | 2 | 2 | 2 | 1
  LYM, Above (pre-vacc) - Above (Month 7) | 3 | 0 | 1 | 1 | 1 | 0 | 1
  LYM, Below (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 1 | 3
  LYM, Below (pre-vacc) - Normal (Month 2) | 2 | 1 | 1 | 0 | 1 | 1 | 3
  LYM, Below (pre-vacc) - Below (Month 2): number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 1 | 3
  LYM, Below (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 1 | 0 | 0 | 0
  LYM, Below (pre-vacc) - Above (Month 2): number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 1 | 3
  LYM, Below (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYM, Below (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 1 | 3
  LYM, Below (pre-vacc) - Normal (Month 7) | 1 | 1 | 1 | 0 | 1 | 1 | 3
  LYM, Below (pre-vacc) - Below (Month 7): number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 1 | 3
  LYM, Below (pre-vacc) - Below (Month 7) | 1 | 0 | 0 | 1 | 0 | 0 | 0
  LYM, Below (pre-vacc) - Above (Month 7): number analyzed (Participants) | 2 | 1 | 1 | 1 | 1 | 1 | 3
  LYM, Below (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MONO, Normal (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 76 | 38 | 39 | 37 | 41 | 44 | 42
  MONO, Normal (pre-vacc) - Normal (Month 2) | 68 | 34 | 36 | 31 | 36 | 40 | 37
  MONO, Normal (pre-vacc) - Below (Month 2): number analyzed (Participants) | 76 | 38 | 39 | 37 | 41 | 44 | 42
  MONO, Normal (pre-vacc) - Below (Month 2) | 6 | 3 | 3 | 4 | 3 | 2 | 5
  MONO, Normal (pre-vacc) - Above (Month 2): number analyzed (Participants) | 76 | 38 | 39 | 37 | 41 | 44 | 42
  MONO, Normal (pre-vacc) - Above (Month 2) | 1 | 1 | 0 | 2 | 1 | 2 | 0
  MONO, Normal (pre-vacc) - Missing (Month 2): number analyzed (Participants) | 76 | 38 | 39 | 37 | 41 | 44 | 42
  MONO, Normal (pre-vacc) - Missing (Month 2) | 1 | 0 | 0 | 0 | 1 | 0 | 0
  MONO, Normal (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 73 | 38 | 38 | 37 | 41 | 39 | 41
  MONO, Normal (pre-vacc) - Normal (Month 7) | 69 | 35 | 34 | 32 | 35 | 35 | 39
  MONO, Normal (pre-vacc) - Below (Month 7): number analyzed (Participants) | 73 | 38 | 38 | 37 | 41 | 39 | 41
  MONO, Normal (pre-vacc) - Below (Month 7) | 3 | 0 | 4 | 2 | 4 | 3 | 1
  MONO, Normal (pre-vacc) - Above (Month 7): number analyzed (Participants) | 73 | 38 | 38 | 37 | 41 | 39 | 41
  MONO, Normal (pre-vacc) - Above (Month 7) | 0 | 2 | 0 | 3 | 2 | 1 | 1
  MONO, Normal (pre-vacc) - Missing (Month 7): number analyzed (Participants) | 73 | 38 | 38 | 37 | 41 | 39 | 41
  MONO, Normal (pre-vacc) - Missing (Month 7) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  MONO, Above (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 1 | 1 | 3 | 1 | 0 | 1 | 1
  MONO, Above (pre-vacc) - Normal (Month 2) | 0 | 1 | 3 | 0 | 0 | 0 | 0
  MONO, Above (pre-vacc) - Below (Month 2): number analyzed (Participants) | 1 | 1 | 3 | 1 | 0 | 1 | 1
  MONO, Above (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MONO, Above (pre-vacc) - Above (Month 2): number analyzed (Participants) | 1 | 1 | 3 | 1 | 0 | 1 | 1
  MONO, Above (pre-vacc) - Above (Month 2) | 1 | 0 | 0 | 1 | 0 | 1 | 1
  MONO, Above (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 1 | 1 | 3 | 1 | 0 | 1 | 1
  MONO, Above (pre-vacc) - Normal (Month 7) | 1 | 1 | 3 | 0 | 0 | 0 | 0
  MONO, Above (pre-vacc) - Below (Month 7): number analyzed (Participants) | 1 | 1 | 3 | 1 | 0 | 1 | 1
  MONO, Above (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MONO, Above (pre-vacc) - Above (Month 7): number analyzed (Participants) | 1 | 1 | 3 | 1 | 0 | 1 | 1
  MONO, Above (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 1 | 0 | 1 | 1
  MONO, Below (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 3 | 4 | 0 | 4 | 3 | 3 | 3
  MONO, Below (pre-vacc) - Normal (Month 2) | 1 | 2 | 0 | 4 | 2 | 1 | 1
  MONO, Below (pre-vacc) - Below (Month 2): number analyzed (Participants) | 3 | 4 | 0 | 4 | 3 | 3 | 3
  MONO, Below (pre-vacc) - Below (Month 2) | 2 | 2 | 0 | 0 | 1 | 2 | 2
  MONO, Below (pre-vacc) - Above (Month 2): number analyzed (Participants) | 3 | 4 | 0 | 4 | 3 | 3 | 3
  MONO, Below (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  MONO, Below (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 3 | 3 | 0 | 4 | 2 | 3 | 3
  MONO, Below (pre-vacc) - Normal (Month 7) | 1 | 2 | 0 | 3 | 2 | 2 | 2
  MONO, Below (pre-vacc) - Below (Month 7): number analyzed (Participants) | 3 | 3 | 0 | 4 | 2 | 3 | 3
  MONO, Below (pre-vacc) - Below (Month 7) | 2 | 1 | 0 | 1 | 0 | 1 | 1
  MONO, Below (pre-vacc) - Above (Month 7): number analyzed (Participants) | 3 | 3 | 0 | 4 | 2 | 3 | 3
  MONO, Below (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Normal (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 74 | 40 | 40 | 40 | 42 | 45 | 42
  NEU, Normal (pre-vacc) - Normal (Month 2) | 63 | 39 | 39 | 36 | 40 | 42 | 41
  NEU, Normal (pre-vacc) - Below (Month 2): number analyzed (Participants) | 74 | 40 | 40 | 40 | 42 | 45 | 42
  NEU, Normal (pre-vacc) - Below (Month 2) | 7 | 1 | 0 | 3 | 1 | 3 | 1
  NEU, Normal (pre-vacc) - Above (Month 2): number analyzed (Participants) | 74 | 40 | 40 | 40 | 42 | 45 | 42
  NEU, Normal (pre-vacc) - Above (Month 2) | 3 | 0 | 1 | 1 | 0 | 0 | 0
  NEU, Normal (pre-vacc) - Missing (Month 2): number analyzed (Participants) | 74 | 40 | 40 | 40 | 42 | 45 | 42
  NEU, Normal (pre-vacc) - Missing (Month 2) | 1 | 0 | 0 | 0 | 1 | 0 | 0
  NEU, Normal (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 72 | 39 | 39 | 40 | 41 | 40 | 41
  NEU, Normal (pre-vacc) - Normal (Month 7) | 69 | 35 | 38 | 37 | 40 | 38 | 39
  NEU, Normal (pre-vacc) - Below (Month 7): number analyzed (Participants) | 72 | 39 | 39 | 40 | 41 | 40 | 41
  NEU, Normal (pre-vacc) - Below (Month 7) | 2 | 3 | 0 | 3 | 1 | 0 | 1
  NEU, Normal (pre-vacc) - Above (Month 7): number analyzed (Participants) | 72 | 39 | 39 | 40 | 41 | 40 | 41
  NEU, Normal (pre-vacc) - Above (Month 7) | 0 | 0 | 1 | 0 | 0 | 2 | 1
  NEU, Normal (pre-vacc) - Missing (Month 7): number analyzed (Participants) | 72 | 39 | 39 | 40 | 41 | 40 | 41
  NEU, Normal (pre-vacc) - Missing (Month 7) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  NEU, Above (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 3 | 2 | 2 | 1 | 1 | 3 | 3
  NEU, Above (pre-vacc) - Normal (Month 2) | 3 | 2 | 2 | 1 | 1 | 3 | 3
  NEU, Above (pre-vacc) - Below (Month 2): number analyzed (Participants) | 3 | 2 | 2 | 1 | 1 | 3 | 3
  NEU, Above (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Above (pre-vacc) - Above (Month 2): number analyzed (Participants) | 3 | 2 | 2 | 1 | 1 | 3 | 3
  NEU, Above (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Above (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 2 | 2 | 2 | 1 | 1 | 3 | 3
  NEU, Above (pre-vacc) - Normal (Month 7) | 2 | 2 | 2 | 1 | 1 | 3 | 3
  NEU, Above (pre-vacc) - Below (Month 7): number analyzed (Participants) | 2 | 2 | 2 | 1 | 1 | 3 | 3
  NEU, Above (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Above (pre-vacc) - Above (Month 7): number analyzed (Participants) | 2 | 2 | 2 | 1 | 1 | 3 | 3
  NEU, Above (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Below (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 3 | 1 | 0 | 1 | 1 | 0 | 1
  NEU, Below (pre-vacc) - Normal (Month 2) | 2 | 1 | 0 | 1 | 1 | 0 | 1
  NEU, Below (pre-vacc) - Below (Month 2): number analyzed (Participants) | 3 | 1 | 0 | 1 | 1 | 0 | 1
  NEU, Below (pre-vacc) - Below (Month 2) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Below (pre-vacc) - Above (Month 2): number analyzed (Participants) | 3 | 1 | 0 | 1 | 1 | 0 | 1
  NEU, Below (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NEU, Below (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 3 | 1 | 0 | 1 | 1 | 0 | 1
  NEU, Below (pre-vacc) - Normal (Month 7) | 1 | 1 | 0 | 1 | 1 | 0 | 0
  NEU, Below (pre-vacc) - Below (Month 7): number analyzed (Participants) | 3 | 1 | 0 | 1 | 1 | 0 | 1
  NEU, Below (pre-vacc) - Below (Month 7) | 2 | 0 | 0 | 0 | 0 | 0 | 1
  NEU, Below (pre-vacc) - Above (Month 7): number analyzed (Participants) | 3 | 1 | 0 | 1 | 1 | 0 | 1
  NEU, Below (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Normal (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 75 | 44 | 41 | 41 | 45 | 46 | 43
  PLA, Normal (pre-vacc) - Normal (Month 2) | 74 | 43 | 40 | 41 | 43 | 46 | 43
  PLA, Normal (pre-vacc) - Below (Month 2): number analyzed (Participants) | 75 | 44 | 41 | 41 | 45 | 46 | 43
  PLA, Normal (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Normal (pre-vacc) - Above (Month 2): number analyzed (Participants) | 75 | 44 | 41 | 41 | 45 | 46 | 43
  PLA, Normal (pre-vacc) - Above (Month 2) | 1 | 1 | 1 | 0 | 1 | 0 | 0
  PLA, Normal (pre-vacc) - Missing (Month 2): number analyzed (Participants) | 75 | 44 | 41 | 41 | 45 | 46 | 43
  PLA, Normal (pre-vacc) - Missing (Month 2) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  PLA, Normal (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 73 | 43 | 40 | 41 | 44 | 41 | 42
  PLA, Normal (pre-vacc) - Normal (Month 7) | 70 | 42 | 39 | 41 | 43 | 40 | 42
  PLA, Normal (pre-vacc) - Below (Month 7): number analyzed (Participants) | 73 | 43 | 40 | 41 | 44 | 41 | 42
  PLA, Normal (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Normal (pre-vacc) - Above (Month 7): number analyzed (Participants) | 73 | 43 | 40 | 41 | 44 | 41 | 42
  PLA, Normal (pre-vacc) - Above (Month 7) | 3 | 0 | 1 | 0 | 1 | 1 | 0
  PLA, Normal (pre-vacc) - Missing (Month 7): number analyzed (Participants) | 73 | 43 | 40 | 41 | 44 | 41 | 42
  PLA, Normal (pre-vacc) - Missing (Month 7) | 0 | 1 | 0 | 0 | 0 | 0 | 0
  PLA, Above (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 7 | 2 | 1 | 4 | 1 | 4 | 3
  PLA, Above (pre-vacc) - Normal (Month 2) | 4 | 2 | 1 | 2 | 0 | 2 | 3
  PLA, Above (pre-vacc) - Below (Month 2): number analyzed (Participants) | 7 | 2 | 1 | 4 | 1 | 4 | 3
  PLA, Above (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Above (pre-vacc) - Above (Month 2): number analyzed (Participants) | 7 | 2 | 1 | 4 | 1 | 4 | 3
  PLA, Above (pre-vacc) - Above (Month 2) | 3 | 0 | 0 | 2 | 1 | 2 | 0
  PLA, Above (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 6 | 2 | 1 | 4 | 1 | 4 | 3
  PLA, Above (pre-vacc) - Normal (Month 7) | 1 | 1 | 0 | 2 | 0 | 1 | 2
  PLA, Above (pre-vacc) - Below (Month 7): number analyzed (Participants) | 6 | 2 | 1 | 4 | 1 | 4 | 3
  PLA, Above (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Above (pre-vacc) - Above (Month 7): number analyzed (Participants) | 6 | 2 | 1 | 4 | 1 | 4 | 3
  PLA, Above (pre-vacc) - Above (Month 7) | 5 | 1 | 1 | 2 | 1 | 3 | 1
  PLA, Below (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0 | 0
  PLA, Below (pre-vacc) - Normal (Month 2) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Below (pre-vacc) - Below (Month 2): number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0 | 0
  PLA, Below (pre-vacc) - Below (Month 2) | 0 | 0 | 1 | 0 | 0 | 0 | 0
  PLA, Below (pre-vacc) - Above (Month 2): number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0 | 0
  PLA, Below (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Below (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0 | 0
  PLA, Below (pre-vacc) - Normal (Month 7) | 1 | 0 | 1 | 0 | 0 | 0 | 0
  PLA, Below (pre-vacc) - Below (Month 7): number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0 | 0
  PLA, Below (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, Below (pre-vacc) - Above (Month 7): number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0 | 0
  PLA, Below (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC, Normal (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 83 | 42 | 42 | 41 | 44 | 49 | 43
  RBC, Normal (pre-vacc) - Normal (Month 2) | 83 | 41 | 42 | 41 | 41 | 47 | 41
  RBC, Normal (pre-vacc) - Below (Month 2): number analyzed (Participants) | 83 | 42 | 42 | 41 | 44 | 49 | 43
  RBC, Normal (pre-vacc) - Below (Month 2) | 0 | 1 | 0 | 0 | 2 | 2 | 1
  RBC, Normal (pre-vacc) - Above (Month 2): number analyzed (Participants) | 83 | 42 | 42 | 41 | 44 | 49 | 43
  RBC, Normal (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  RBC, Normal (pre-vacc) - Missing (Month 2): number analyzed (Participants) | 83 | 42 | 42 | 41 | 44 | 49 | 43
  RBC, Normal (pre-vacc) - Missing (Month 2) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  RBC, Normal (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 80 | 42 | 41 | 41 | 43 | 44 | 42
  RBC, Normal (pre-vacc) - Normal (Month 7) | 78 | 42 | 41 | 41 | 41 | 43 | 42
  RBC, Normal (pre-vacc) - Below (Month 7): number analyzed (Participants) | 80 | 42 | 41 | 41 | 43 | 44 | 42
  RBC, Normal (pre-vacc) - Below (Month 7) | 1 | 0 | 0 | 0 | 1 | 1 | 0
  RBC, Normal (pre-vacc) - Above (Month 7): number analyzed (Participants) | 80 | 42 | 41 | 41 | 43 | 44 | 42
  RBC, Normal (pre-vacc) - Above (Month 7) | 1 | 0 | 0 | 0 | 1 | 0 | 0
  RBC, Above (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 0 | 1
  RBC, Above (pre-vacc) - Normal (Month 2) | 0 | 2 | 0 | 0 | 0 | 0 | 1
  RBC, Above (pre-vacc) - Below (Month 2): number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 0 | 1
  RBC, Above (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC, Above (pre-vacc) - Above (Month 2): number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 0 | 1
  RBC, Above (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC, Above (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 0 | 1
  RBC, Above (pre-vacc) - Normal (Month 7) | 0 | 2 | 0 | 0 | 0 | 0 | 1
  RBC, Above (pre-vacc) - Below (Month 7): number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 0 | 1
  RBC, Above (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC, Above (pre-vacc) - Above (Month 7): number analyzed (Participants) | 0 | 2 | 0 | 0 | 0 | 0 | 1
  RBC, Above (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC, Below (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 0 | 2 | 1 | 4 | 2 | 1 | 2
  RBC, Below (pre-vacc) - Normal (Month 2) | 0 | 1 | 0 | 4 | 2 | 1 | 1
  RBC, Below (pre-vacc) - Below (Month 2): number analyzed (Participants) | 0 | 2 | 1 | 4 | 2 | 1 | 2
  RBC, Below (pre-vacc) - Below (Month 2) | 0 | 1 | 1 | 0 | 0 | 0 | 1
  RBC, Below (pre-vacc) - Above (Month 2): number analyzed (Participants) | 0 | 2 | 1 | 4 | 2 | 1 | 2
  RBC, Below (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  RBC, Below (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 0 | 1 | 1 | 4 | 2 | 1 | 2
  RBC, Below (pre-vacc) - Normal (Month 7) | 0 | 1 | 1 | 2 | 2 | 1 | 1
  RBC, Below (pre-vacc) - Below (Month 7): number analyzed (Participants) | 0 | 1 | 1 | 4 | 2 | 1 | 2
  RBC, Below (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 2 | 0 | 0 | 1
  RBC, Below (pre-vacc) - Above (Month 7): number analyzed (Participants) | 0 | 1 | 1 | 4 | 2 | 1 | 2
  RBC, Below (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC, Normal (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 74 | 39 | 41 | 41 | 42 | 45 | 41
  WBC, Normal (pre-vacc) - Normal (Month 2) | 71 | 37 | 39 | 40 | 41 | 42 | 40
  WBC, Normal (pre-vacc) - Below (Month 2): number analyzed (Participants) | 74 | 39 | 41 | 41 | 42 | 45 | 41
  WBC, Normal (pre-vacc) - Below (Month 2) | 1 | 1 | 0 | 0 | 0 | 2 | 1
  WBC, Normal (pre-vacc) - Above (Month 2): number analyzed (Participants) | 74 | 39 | 41 | 41 | 42 | 45 | 41
  WBC, Normal (pre-vacc) - Above (Month 2) | 2 | 1 | 2 | 1 | 0 | 1 | 0
  WBC, Normal (pre-vacc) - Missing (Month 2): number analyzed (Participants) | 74 | 39 | 41 | 41 | 42 | 45 | 41
  WBC, Normal (pre-vacc) - Missing (Month 2) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  WBC, Normal (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 71 | 38 | 40 | 41 | 41 | 40 | 40
  WBC, Normal (pre-vacc) - Normal (Month 7) | 69 | 36 | 38 | 41 | 38 | 37 | 37
  WBC, Normal (pre-vacc) - Below (Month 7): number analyzed (Participants) | 71 | 38 | 40 | 41 | 41 | 40 | 40
  WBC, Normal (pre-vacc) - Below (Month 7) | 0 | 1 | 1 | 0 | 2 | 1 | 1
  WBC, Normal (pre-vacc) - Above (Month 7): number analyzed (Participants) | 71 | 38 | 40 | 41 | 41 | 40 | 40
  WBC, Normal (pre-vacc) - Above (Month 7) | 1 | 0 | 1 | 0 | 1 | 2 | 2
  WBC, Normal (pre-vacc) - Missing (Month 7): number analyzed (Participants) | 71 | 38 | 40 | 41 | 41 | 40 | 40
  WBC, Normal (pre-vacc) - Missing (Month 7) | 1 | 1 | 0 | 0 | 0 | 0 | 0
  WBC, Above (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 4 | 7 | 2 | 2 | 2 | 5 | 4
  WBC, Above (pre-vacc) - Normal (Month 2) | 3 | 6 | 2 | 1 | 2 | 2 | 4
  WBC, Above (pre-vacc) - Below (Month 2): number analyzed (Participants) | 4 | 7 | 2 | 2 | 2 | 5 | 4
  WBC, Above (pre-vacc) - Below (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC, Above (pre-vacc) - Above (Month 2): number analyzed (Participants) | 4 | 7 | 2 | 2 | 2 | 5 | 4
  WBC, Above (pre-vacc) - Above (Month 2) | 1 | 1 | 0 | 1 | 0 | 3 | 0
  WBC, Above (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 4 | 7 | 2 | 2 | 2 | 5 | 4
  WBC, Above (pre-vacc) - Normal (Month 7) | 3 | 6 | 1 | 2 | 2 | 3 | 4
  WBC, Above (pre-vacc) - Below (Month 7): number analyzed (Participants) | 4 | 7 | 2 | 2 | 2 | 5 | 4
  WBC, Above (pre-vacc) - Below (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC, Above (pre-vacc) - Above (Month 7): number analyzed (Participants) | 4 | 7 | 2 | 2 | 2 | 5 | 4
  WBC, Above (pre-vacc) - Above (Month 7) | 1 | 1 | 1 | 0 | 0 | 2 | 0
  WBC, Below (pre-vacc) - Normal (Month 2): number analyzed (Participants) | 5 | 0 | 0 | 2 | 2 | 0 | 1
  WBC, Below (pre-vacc) - Normal (Month 2) | 4 | 0 | 0 | 2 | 2 | 0 | 1
  WBC, Below (pre-vacc) - Below (Month 2): number analyzed (Participants) | 5 | 0 | 0 | 2 | 2 | 0 | 1
  WBC, Below (pre-vacc) - Below (Month 2) | 1 | 0 | 0 | 0 | 0 | 0 | 0
  WBC, Below (pre-vacc) - Above (Month 2): number analyzed (Participants) | 5 | 0 | 0 | 2 | 2 | 0 | 1
  WBC, Below (pre-vacc) - Above (Month 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  WBC, Below (pre-vacc) - Normal (Month 7): number analyzed (Participants) | 5 | 0 | 0 | 2 | 2 | 0 | 1
  WBC, Below (pre-vacc) - Normal (Month 7) | 3 | 0 | 0 | 0 | 2 | 0 | 1
  WBC, Below (pre-vacc) - Below (Month 7): number analyzed (Participants) | 5 | 0 | 0 | 2 | 2 | 0 | 1
  WBC, Below (pre-vacc) - Below (Month 7) | 2 | 0 | 0 | 2 | 0 | 0 | 0
  WBC, Below (pre-vacc) - Above (Month 7): number analyzed (Participants) | 5 | 0 | 0 | 2 | 2 | 0 | 1
  WBC, Below (pre-vacc) - Above (Month 7) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs: During the 7-day period after each vaccination. Unsolicited AEs: During the 30-day period after vaccination. SAEs: From Day 0 up to Month 12.
Description: The Total Number of Participants Affected by Other AEs was analyzed separately for solicited AEs and unsolicited AEs. An analysis of all AEs was not possible, and the relevant data are no longer available. The Total Number of Participants Affected in Other AEs table is populated with the highest number of participants affected in the Other AEs table.
Arm/Group | HPV-16/18 Group | HPV-TETRA A Group | HPV-TETRA B Group | HPV-TETRA C Group | HPV-TETRA D Group | HPV-TETRA E Group | HPV-TETRA F Group
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/50 | 0/49 | 0/48 | 0/48 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 2/88 | 2/50 | 1/49 | 3/48 | 2/48 | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 81/88 | 48/50 | 46/49 | 45/48 | 44/48 | 50/50 | 47/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HPV-16/18 Group (N=88) | HPV-TETRA A Group (N=50) | HPV-TETRA B Group (N=49) | HPV-TETRA C Group (N=48) | HPV-TETRA D Group (N=48) | HPV-TETRA E Group (N=50) | HPV-TETRA F Group (N=50)
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myelitis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | HPV-16/18 Group (N=88) | HPV-TETRA A Group (N=50) | HPV-TETRA B Group (N=49) | HPV-TETRA C Group (N=48) | HPV-TETRA D Group (N=48) | HPV-TETRA E Group (N=50) | HPV-TETRA F Group (N=50)
Pain* (General disorders) | 81/86 | 48/49 | 46/47 | 45/46 | 44/46 | 50 | 47/48 — *Solicited symptom during the 7-day post-vaccination period (across doses)
Redness* (General disorders) | 36/86 | 28/49 | 15/47 | 22/46 | 24/46 | 22 | 25/48 — *Solicited symptom during the 7-day post-vaccination period (across doses)
Swelling* (General disorders) | 33/86 | 22/49 | 12/47 | 18/46 | 21/46 | 27 | 19/48 — *Solicited symptom during the 7-day post-vaccination period (across doses)
Arthralgia* (General disorders) | 11/86 | 13/49 | 9/47 | 11/46 | 11/46 | 9 | 11/48 — *Solicited symptom during the 7-day post-vaccination period (across doses)
Fatigue* (General disorders) | 54/86 | 33/49 | 30/47 | 32/46 | 25/46 | 34 | 31/48 — *Solicited symptom during the 7-day post-vaccination period (across doses)
Fever* (General disorders) | 10/86 | 4/49 | 4/47 | 3/46 | 9/46 | 4 | 2/48 — *Solicited symptom during the 7-day post-vaccination period (across doses)
Gastrointestinal* (General disorders) | 36/86 | 15/49 | 18/47 | 20/46 | 17/46 | 17 | 18/48 — *Solicited symptom during the 7-day post-vaccination period (across doses)
Headache (solicited)* (General disorders) | 45/86 | 24/49 | 23/47 | 31/46 | 22/46 | 33 | 27/48 — *Solicited symptom during the 7-day post-vaccination period (across doses)
Myalgia* (General disorders) | 25/86 | 18/49 | 19/47 | 16/46 | 17/46 | 19 | 15/48 — *Solicited symptom during the 7-day post-vaccination period (across doses)
Rash* (General disorders) | 6/86 | 4/49 | 2/47 | 2/46 | 4/46 | 3 | 2/48 — *Solicited symptom during the 7-day post-vaccination period (across doses)
Urticaria* (General disorders) | 3/86 | 2/49 | 3/47 | 0/46 | 0/46 | 1 | 3/48 — *Solicited symptom during the 7-day post-vaccination period (across doses)
Diarrhea** (Gastrointestinal disorders) | 3 | 1 | 1 | 4 | 3 | 0 | 0 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)
Nausea** (Gastrointestinal disorders) | 3 | 3 | 1 | 3 | 0 | 0 | 1 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)
Toothache** (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 4 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)
Injection site pruritus** (General disorders) | 1 | 3 | 0 | 1 | 0 | 0 | 0 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)
Injection site reaction** (General disorders) | 1 | 3 | 1 | 1 | 1 | 1 | 2 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)
Cystitis** (Infections and infestations) | 1 | 1 | 3 | 0 | 1 | 2 | 0 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)
Influenza** (Infections and infestations) | 0 | 0 | 0 | 1 | 3 | 0 | 3 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)
Nasopharyngitis** (Infections and infestations) | 9 | 3 | 5 | 2 | 3 | 5 | 6 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)
Upper respiratory tract infection** (Infections and infestations) | 4 | 4 | 9 | 4 | 6 | 7 | 5 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)
Dizziness** (Nervous system disorders) | 2 | 3 | 1 | 1 | 0 | 1 | 2 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)
Headache (unsolicited)** (Nervous system disorders) | 13 | 8 | 7 | 4 | 7 | 5 | 6 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)
Dysmenorhoea** (Reproductive system and breast disorders) | 1 | 3 | 3 | 1 | 2 | 1 | 0 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)
Pharyngolaryngeal Pain** (Respiratory, thoracic and mediastinal disorders) | 11 | 1 | 2 | 0 | 3 | 4 | 4 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)
Rhinitis** (Infections and infestations) | 3 | 0 | 1 | 0 | 0 | 0 | 3 — **Unsolicited symptom during the 30-day post-vaccination period (across doses)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial